CLINICAL TRIAL: NCT02313610
Title: Efficacy and Safety of Qinbudan as an Adjunct Therapy in Patients Receiving Standard Combination Therapy for Retreatment Pulmonary Tuberculosis: A Randomized, Double-blind, Placebo-controlled Multicenter Clinical Trial
Brief Title: Efficacy and Safety of Qinbudan as an Adjunct Therapy for Retreatment Pulmonary Tuberculosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DS11036
Record Dates: First submitted 2014-12-07; First posted 2014-12-10 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2014-12

CONDITIONS: Pulmonary Tuberculosis
Keywords: Retreatment Pulmonary Tuberculosis, Qinbudan,
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Qinbudan (Experimental): the patient will receive 2HRZES/6HRE follow guidelines of the implementation of China tuberculosis control program （2HRZES/6HRE means： Intensive phase: isoniazid（H）, rifampicin（R）, pyrazinamide（Z）, ethambutol（E）, streptomycin（S）, once, for two months（2）；Consolidation: isoniazid（H）, rifampicin（R）, ethambutol（E）, once, for six months（6）.） Intervention: Qinbudan table, table, 4, thrice a day, 8 months
  Interventions: Drug: Qinbudan
- Control Qinbudan Placebo (Placebo Comparator): the patient will receive 2HRZES/6HRE follow guidelines of the implementation of China tuberculosis control program（2HRZES/6HRE means： Intensive phase: isoniazid（H）, rifampicin（R）, pyrazinamide（Z）, ethambutol（E）, streptomycin（S）, once, for two months（2）；Consolidation: isoniazid（H）, rifampicin（R）, ethambutol（E）, once, for six months（6）.） Intervention: Qinbudan Placebo, table, 4, thrice a day, 8 months
  Interventions: Drug: Qinbudan Placebo

INTERVENTIONS:
Drug: Qinbudan — Contains three kinds of traditional Chinese medicine radix scutellariae, radix stemona, liquorice
  Other Names: Qinbudan table
  Arms: Qinbudan
Drug: Qinbudan Placebo — Qinbudan Placebo was the same as therapeutic drug in package,shape,size.
  Other Names: Qinbudan table Placebo
  Arms: Control Qinbudan Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Chinese medicine Qinbudan in Patients Receiving Standard Combination Therapy for Retreatment Pulmonary Tuberculosis.

DETAILED DESCRIPTION:
Retreatment of tuberculosis involves the management of entities as diverse as relapse, failure, treatment after default, and poor patient adherence to the previous treatment. The emergence of conditions for selection of resistance (failure and partial abandonment) is a matter of great concern. The current chemotherapy is the primary interventions, but the long-term drug combination therapy often leads to adverse reactions. The purpose of this study that is to exploring the role of Chinese medicine Qinbudan on Patients who are initially sputum smear positive or culture-positive who have been treated previously for pulmonary tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are initially sputum smear positive (at least two smears as "1+" or at least have a smear as "2+" and above) or culture-positive for pulmonary tuberculosis who have been treated previously
* Aged 18 -65 years of age
* Patients who are willing to give written informed consent

Exclusion Criteria:

* Participation in another clinical trial 1 month prior to study entry
* Female patients in lactation period, pregnancy or planning to get pregnant during the trial
* Patients who are allergic to the therapeutic medicine
* Patients with severe primary diseases such as cancer, cardiovascular system, digestive system, kidney and hematopoietic system diseases
* Patients co-infected with HIV, hepatitis B or hepatitis C
* Patients with mental illness, acrasia
* Abnormal liver function or combined with other underlying liver disease (fatty liver, alcoholic liver)
* Patients with diabetes, Plasma glucose poorly controlled undertaking
* Patients with auditory dysfunction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2011-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
The time of sputum conversion between the 2 groups will be evaluated | Measured during the 8 months treatment period

SECONDARY OUTCOMES:
Time to resolution of all pulmonary tuberculosis symptoms | 8 months
Resolution of chest X-ray changes of patients | 8 months to baseline
T cell classification in peripheral blood | 8 months to baseline
  immunologic function(CD3、CD4、CD8)
Erythrocyte Sedimentation Rata | once every month during the 8 months treatment period
The cure rate will be evaluated as the primary parameter of efficacy | 8-9 months
The relapse in patients of both groups will be compared | at 12 months after the completion of the therapy

CONTACTS AND LOCATIONS:
Overall Officials: Guang Ji, Study Chair — Shanghai University of Traditional Chinese Medicine
Locations (12):
- China (12):
  - Hebei provincial chest hospital, Shijiazhuang, Hebei
  - The first affiliated hospital of Xinxiang Medical University, Xinxiang, Henan
  - Wuhan tuberculosis dispensary, Wuhan, Hubei
  - Jiangxi provincial chest hospital, Nanchang, Jiangxi
  - Shenyang chest hospital, Shenyang, Liaoning
  - Uygur Autonomous Region of Xinjiang Chest Hospital, Ürümqi, Xinjiang
  - Beijing chest hospital,Capital medical university, Beijing
  - The first affiliated hospital of chongqing medical university, Chongqing
  - The 85th hospital of chinese people's liberation army, Shanghai
  - Shanghai pulmonary hospital affiliated Tongji University, Shanghai
  - Shenzhen Donghu hospital, Shenzhen
  - Tianjin Haihe hospital, Tianjin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang SY, Fu JY, Guo XY, Wu DZ, Zhang T, Li C, Qiu L, Shao CR, Xiao HP, Chu NH, Deng QY, Zhang X, Yan XF, Wang ZL, Zhang ZJ, Jiang X, Zheng YJ, Zheng PY, Zhang HY, Lu ZH. Improvement cues of lesion absorption using the adjuvant therapy of traditional Chinese medicine Qinbudan tablet for retreatment pulmonary tuberculosis with standard anti-tuberculosis regimen. Infect Dis Poverty. 2020 May 7;9(1):50. doi: 10.1186/s40249-020-00660-z. PMID 32381098